CLINICAL TRIAL: NCT07107776
Title: Central Venous Oxygen Saturation Impact on Prognosis of Post Arrest Patients
Brief Title: Central Venous Oxygen Saturation Prognostic Impact in Post Arrest Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lydia Mamdouh Sadek Botros, Doctor and master student in critical care medicine l, Assiut University
Other Study IDs: CVO2 prognosis in post arrest
Record Dates: First submitted 2025-07-29; First posted 2025-08-06 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Post Arrest Patients
Keywords: post arrest patients; central venous oxygen saturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — central venous blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aim will be to assess the prognostic impact and value of central venous oxygen saturation on post arrest patients.

DETAILED DESCRIPTION:
Central venous oxygen saturation (ScvO₂) is a very important measurement which can be easily taken in a critical care environment by both medical and nursing staff. It provides an understanding of the patient's oxygen delivery, oxygen consumption and cardiac output. It has a key role within early goal-directed therapy and has been shown to decrease mortality when taken and analysed appropriately. (Central venous oxygen saturation: analysis, clinical use and effects on mortality,2013) Venous oxygen saturation (SvO2) measures the blood's oxygen content returning to the right side of the heart after perfusing the entire body. When the oxygen supply is insufficient to meet the metabolic demands of the tissues, an abnormal SvO2 ensues and reflects an inadequacy in systemic oxygenation. SvO2 is, therefore, dependent on oxygen delivery and oxygen extraction. Venous oximetry is used in specific clinical settings of hemodynamic instability, such as in critical illnesses, perioperative periods of major surgeries, heart failure, sepsis andd post arrest patients. The venous blood in the pulmonary artery represents oxygen extraction in the whole body and is called mixed venous oxygen saturation (SmvO2). It was measured using a pulmonary artery catheter (PAC). A second, less invasive method of measuring SvO2 is via a central venous catheter (CVC) positioned in the superior vena cava and is called the central venous oxygen saturation (ScvO2).

Central venous oxygen saturation (ScvO(2)) is suggested to reflect the adequacy of oxygen delivery, and the main objective of the present study was to determine whether ScvO(2) is associated with outcome in haemodynamically stabilized post arrest patients predicting mortality and outcome based on central venous oxygen saturation

ELIGIBILITY:
Inclusion Criteria:

* adults above 16 years old, critically ill patients
* both genders
* post arrest patients

Exclusion Criteria:

* if patients does not experience cardiac arrest

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: post arrest patients in assiut university hospital both genders above 16 years old
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
central venous oxygen saturation impact on prognosis of post arrest patients | time of follow up expected from time of successful ROSC until full improvement or recurrent arrest and death From date of cardiac arrest until date of first documented improvement or date of death due to any cause whichever came first assessed up in 2 mo
  evaluating prognostic impact of oxygen saturation extracted from a central venous line blood sample on post arrest patients sample from (internal jagular vein) more or less than 50% oxygen saturation on prognosis of post arrest patients and recurrent arrests and overall improvement and time of expected and full recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gallet R, Lellouche N, Mitchell-Heggs L, Bouhemad B, Bensaid A, Dubois-Rande JL, Gueret P, Lim P. Prognosis value of central venous oxygen saturation in acute decompensated heart failure. Arch Cardiovasc Dis. 2012 Jan;105(1):5-12. doi: 10.1016/j.acvd.2011.10.005. Epub 2012 Jan 13. PMID 22369912
- [Background] Grand J, Hassager C, Schmidt H, Molstrom S, Nyholm B, Hoigaard HF, Dahl JS, Meyer M, Beske RP, Obling L, Kjaergaard J, Moller JE. Serial assessments of cardiac output and mixed venous oxygen saturation in comatose patients after out-of-hospital cardiac arrest. Crit Care. 2023 Oct 27;27(1):410. doi: 10.1186/s13054-023-04704-2. PMID 37891623
- [Background] Rodriguez-Scarpetta MA, Sepulveda-Tobon AM, Daza-Arana JE, Lozada-Ramos H, Alzate-Sanchez RA. Central Oxygen Venous Saturation and Mortality in Patients Undergoing Coronary Artery Bypass Grafting. Ther Clin Risk Manag. 2023 Jun 3;19:447-454. doi: 10.2147/TCRM.S407454. eCollection 2023. PMID 37292584